CLINICAL TRIAL: NCT02546050
Title: Effects of Metformin on Human Gut Microbiota
Brief Title: The Effect of Metformin on Composition of Human Gut Bacteria
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oluf Borbye Pedersen (Other)
Responsible Party: Sponsor-Investigator, Oluf Borbye Pedersen, Director, Professor, dr.med, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NNF-CBMR 2015-000199-86; 2015-000199-86 (EudraCT Number)
Record Dates: First submitted 2015-07-01; First posted 2015-09-10 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Healthy
Keywords: Gut microbiota; metformin; Metabolism; Metagenomics; Metabolomics
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metformin (Experimental): 18 weeks study with intervention during week 6 to 12: the intervention consist of 500 mg of metformin once daily for week 7, then 500 mg twice daily week 8, 1000 mg + 500 mg daily week 9 and 1000 mg + 1000 mg daily for weeks 10-12.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin

SUMMARY:
OBJECTIVE: Investigate structural changes in the human gut microbiota and associated changes in metabolic markers in urine, saliva, blood and fecal samples following metformin treatment.

DESIGN: An, 18 week, one-armed cross over intervention trial consisting of a 6-week pre-intervention period, 6-week intervention period and a 6-week post-intervention period. 25 healthy young men will be included in the trial.

INTERVENTION: Six-week Metformin treatment to young healthy men.

DETAILED DESCRIPTION:
An, 18 weeks, one-armed cross over intervention trial consisting of a 6-weeks pre-intervention period, 6-weeks intervention period and a 6-weeks post-intervention period. 25 healthy young men will be included in the trial. The pre-intervention period is the control period with no treatment. During the intervention period participants will receive 500 mg of metformin once daily the 1st week, then 500 mg twice daily the 2nd week, 1000 mg + 500 mg daily the 3rd week and 1000 mg + 1000 mg daily the remaining three weeks. Post-interventional investigators will examine gut microbiota of the participants 6 weeks after completion of the intervention period.

MESUREMENTS: Altered composition of gut microbiota as investigated by 16S rRNA sequencing is the primary outcome of this study. Secondary outcomes are to investigate changes in metabolic and inflammatory markers in blood and fecal samples. Blood, urine, saliva and fecal samples will be stored for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Male
* HbA1c < 5.7 % (39 mmol/mol)
* Caucasian (self-report of parental ethnicity)
* Weight stabile with 18.5 kg/m2 < BMI < 27.0 kg/m2
* Normal kidney function as evaluated by normal p-creatinine for age

Exclusion Criteria:

* Oral intake of any form of prescribed medication two months prior to recruitment
* Chronic or acute illness
* Previous gastro-intestinal operation excluding appendicitis
* Any other significant medical reason for exclusion as determined by the investigator
* Unable to give informed consent
* Need of medical treatment during the study period

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2015-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Structural changes in the human gut microbiota. | Baseline, 4 , 7, 8, 10, 11 , 13, 16, and 18 weeks
  Fecal samples are collected in order to characterize the gut microbiota composition.
  Microbial DNA will be subjected to sequencing, microbial gene analyses, including taxonomic and functional annotation.

SECONDARY OUTCOMES:
Changes in plasma glucose and HbA1c levels | Baseline and at week 7,10,13 and 18
  Venous blood will be collected. The samples will be analyzed for plasma glucose and HbA1c, and correlated to changes in gut microbiota composition
Changes in insulin metabolism | Baseline and at week 7,10,13 and 18
  Venous blood will be collected. The samples will be analyzed for serum insulin and C-peptide levels. Changes will be correlated to changes in gut microbiota composition.
Changes in inflammatory markers in blood samples. | Baseline and at week 7,10,13 and 18
  Venous blood will be collected. The samples will be analyzed for markers of inflammation such as high sensitive C-reactive protein.
Changes in kidney function tests. | Baseline and at week 7,10,13 and 18
  Venous blood will be collected. The samples will be analyzed for plasma creatinine and correlated to gut microbiota changes
Changes in liver function tests. | Baseline and at week 7,10,13 and 18
  Venous blood will be collected. The samples will be analyzed for liver function test and correlated to gut microbiota changes
Serum Cobalamin | Baseline and at week 7,10,13 and 18
  Venous blood will be collected. The samples will be analyzed for serum cobalamin and correlated to gut microbiota changes
Metformin plasma level | At week 10 and 13.
  Plasma levels of metformin will be measured at visits 3 and 4 in order to test for compliance. Plasma metformin concentrations will be correlated to changes in gut microbiota composition and function
Blood pressure | Baseline and at week 7,13 and 18
  Systolic and diastolic blood pressure are measured in the inclined position after a five minute rest using an automated sphygmomanometer. The measurement is repeated three times. Participants are instructed not to talk during the measurements.
Heart rate | Baseline and at week 7,13 and 18
  Heart rate is measured in the inclined position after a five minute rest using an automated sphygmomanometer. The measurement is repeated three times. Participants are instructed not to talk during the measurements.
Anthropometrics characteristics | Baseline and at week 7,13 and 18
  Weight is measured using standardized procedures.
Anthropometrics characteristics | Baseline and at week 7,13 and 18
  Height is measured using standardized procedures.
Anthropometrics characteristics | Baseline and at week 7,13 and 18
  Waist- and hip circumference are measured using standardized procedures.
Bio-electrical impedance. | Baseline and at week 7,13 and 18
  Body composition will be measured through bio-electrical impedance
GI symptoms | Baseline and at week 7, 10, 13 and 18.
  Changes in gastrointestinal symptoms of participants by validated VAS-questionnaire concerning following parameters: Overall abdominal symptoms, abdominal pain, bloating, flatulence, satisfaction with stool consistence, constipation, diarrhea, tiredness, nausea, metallic taste.

CONTACTS AND LOCATIONS:
Overall Officials: Oluf Pedersen, MD, Professor, Principal Investigator — The Novo Nordisk Foundation Center for Basic Metabolic Research, Faculty of Health and Medical Sciences University of Copenhagen
Locations (1):
- The Novo Nordisk Foundation Center of Basic Metabolic Research, Section for Metabolic Genetics, University of Copenhagen, Copenhagen, Copenhagen Ø, Denmark

REFERENCES:
- [Derived] Bryrup T, Thomsen CW, Kern T, Allin KH, Brandslund I, Jorgensen NR, Vestergaard H, Hansen T, Hansen TH, Pedersen O, Nielsen T. Metformin-induced changes of the gut microbiota in healthy young men: results of a non-blinded, one-armed intervention study. Diabetologia. 2019 Jun;62(6):1024-1035. doi: 10.1007/s00125-019-4848-7. Epub 2019 Mar 23. PMID 30904939